CLINICAL TRIAL: NCT00511004
Title: Effect of Albendazole Dose and Interval on Brugia Malayi Microfilarial Clearance in India: A Randomized, Open Label Study
Brief Title: Effect of Albendazole Dose on Treatment of Lymphatic Filariasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 999907197; 07-I-N197 (Other: NIAID IRB)
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-07

CONDITIONS: Lymphatic Filariasis
Keywords: Brugia Malayi; Lymphatic Filariasis; Albendazole; Diethylcarbamazine
MeSH Terms: conditions — Elephantiasis, Filarial | interventions — Albendazole; Diethylcarbamazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diethylcarbamazine/Albendazole -STD (Active Comparator): Standard therapy of DEC (300mg) and albendazole (400mg) yearly
  Interventions: Drug: Albendazole; Drug: Diethylcarbamazine
- Diethylcarbamazine/Albendazole- HD1 (Active Comparator): High dose of DEC (300mg) and albendazole (800mg) yearly
  Interventions: Drug: Albendazole; Drug: Diethylcarbamazine
- Diethylcarbamazine/Albendazole-HD2 (Active Comparator): High dose of DEC (300mg) and albendazole (800mg) twice yearly (every 6 months)
  Interventions: Drug: Albendazole; Drug: Diethylcarbamazine

INTERVENTIONS:
Drug: Albendazole — Comparing 400 mg to 800 mg dose
  Other Names: Zentel
Drug: Diethylcarbamazine — Providing diethylcarbamazine more frequently in combination with albendazole
  Other Names: Banocide

SUMMARY:
This study is conducted in Kerala, India. It will determine whether a new treatment regimen of albendazole and diethylcarbamazine (DEC) for lymphatic filariasis can eliminate the disease more quickly than the standard regimen. Lymphatic filariasis is caused by infection with very small parasitic worms that are spread by mosquitoes. The disease can cause swelling of the arms, legs, breast and scrotum and can progress to permanent swelling of the legs or arms called elephantiasis. The study will see if a higher and more frequent dose of albendazole is better at clearing filarial worms from the blood than the current treatment.

Healthy people between 18 and 55 years of age who are in good health and who are infected with filarial worms may be eligible for this study.

Participants undergo the following procedures:

3-day hospital stay at the Filariasis Chemotherapy Unit of the T.D. Medical College Hospital in Kerala, India

* Random assignment to receive either: 400 mg albendazole and DEC 300 mg given once a year for 2 years (standard treatment); or 800 mg albendazole and DEC 300 mg given once a year for 2 years; or 800 mg albendazole and DEC 300 mg given twice a year for 2 years.
* Urine pregnancy test for women of childbearing age .
* Ultrasound test to look for filarial worms.
* Treatment dose.
* Monitoring for symptoms

  6-month 3-day hospital stay
* Medical history, physical examination and blood test.
* Repeat ultrasound in subjects whose first ultrasound detected adult worms.
* Treatment dose for subjects receiving medicine every 6 months.
* Urine pregnancy test for women of childbearing age.

  1-year 3-day hospital stay
* Medical history, physical examination and blood test.
* Treatment dose.
* Repeat ultrasound in subjects whose first ultrasound detected adult worms.
* Urine pregnancy test for women of childbearing age.

  18-month 3-day hospital stay
* Medical history, physical examination and blood test.
* Treatment dose for subjects receiving medicine every 6 months.
* Urine pregnancy test for women of childbearing age.

  24-month 3-day hospital stay
* Medical history, physical examination and blood test.
* Treatment dose.
* Repeat ultrasound in subjects whose first ultrasound detected adult worms.
* Urine pregnancy test for women of childbearing age.

DETAILED DESCRIPTION:
Albendazole and diethylcarbamazine (DEC) are currently used in combination for annual mass treatment of lymphatic filariasis in all parts of the world except Africa. Although the drugs have been donated, the cost of such programs is very high and has proven to be a major impediment to the success of programs in many countries with limited financial resources. Data from albendazole treatment of other filarial infections and one study comparing single to multi-dose DEC/albendazole in lymphatic filariasis suggest that increased dose and/or frequency of albendazole dosing may be more effective in clearing microfilariae. In this study, 75 volunteers with microfilaremic Brugia malayi infection will be randomized to receive standard annual therapy (albendazole 400 mg + DEC 300 mg), annual therapy with increased dosing of albendazole (albendazole 800 mg + DEC 300 mg), or semiannual therapy with an increased albendazole dose (albendazole 800 mg + DEC 300 mg). Microfilarial levels will be followed every 6 months for 2 years to determine whether the higher dose, and/or the more frequent regimen, is more effective.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for Screening:

* Age 18 years to 55 years inclusive
* Both genders
* Not pregnant or breastfeeding by history
* If selected, subjects must be willing to spend 3 days on the Filariasis Chemotherapy Unit at the T.D. Medical College Hospital, Alleppey, Kerala, India
* If selected, subjects must be willing to undergo nighttime blood draws once every 6 months and Doppler ultrasound twice yearly for 2 years
* If selected, agree to have blood stored for future studies
* Ability to understand and give informed consent

Inclusion Criteria for Treatment:

* Age 18 to 55 years inclusive
* Men and non-pregnant or non-breast feeding women
* Microfilarial levels greater than 50mf/mL
* Willingness to spend 3 days on the Filariasis Chemotherapy Unit at the T.D. Medical College Hospital, Alleppey, Kerala, India every 6 months for 2 years
* Willingness to undergo nighttime blood draws once every 6 months for 2 years
* Ability to understand and give informed consent
* Hemaglobin (Hgb) levels for inclusion greater than 9 g/dL
* Creatinine (Cr) less than or equal to 1.2 mg/dL
* Alanine aminotransferase (ALT) less than 30 U/L
* Willingness to have blood stored for future studies

EXCLUSION CRITERIA:

Exclusion Criteria for Screening:

* Age less than 18 years or greater than 55 years
* Pregnant or breast feeding by history

Exclusion Criteria for Treatment:

* Non-volunteers
* Age less than 18 years or greater than 55 years
* Pregnant or breast feeding
* Hgb levels less than or equal to 9 g/dL
* Cr greater than 1.3 mg/dL
* ALT greater than 30 U/L
* Alcohol consumption of more than 2 beers or other alcohol-containing drinks/day within a week of each drug administration
* Temperature greater than 37.5 degrees Celsius
* Serious medical illness
* History of benzimidazole allergy
* History of DEC allergy
* Use of albendazole or DEC within past 6 months
* Unwillingness to comply with required study visits

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Nutman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Filariasis Chemotherapy Unit (FCU), T.D. Medical Hospital, Alleppey, Kerala, India

REFERENCES:
- [Background] Edwards G, Awadzi K, Breckenridge AM, Gilles HM, Orme ML, Ward SA. Diethylcarbamazine disposition in patients with onchocerciasis. Clin Pharmacol Ther. 1981 Oct;30(4):551-7. doi: 10.1038/clpt.1981.202. PMID 7285488
- [Background] Taylor HR, Greene BM. Ocular changes with oral and transepidermal diethylcarbamazine therapy of onchocerciasis. Br J Ophthalmol. 1981 Jul;65(7):494-502. doi: 10.1136/bjo.65.7.494. PMID 7020746
- [Background] Partono F, Purnomo, Oemijati S, Soewarta A. The long term effects of repeated diethylcarbamazine administration with special reference to microfilaraemia and elephantiasis. Acta Trop. 1981 Sep;38(3):217-25. PMID 6118029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults living in Kerala, India with Brugia malayi microfilaremia were recruited from field sites around the city of Alleppey and the study performed in the outpatient department of the TD Medical College.
Groups:
- Standard Therapy Annual DEC/ALB: Group randomized to standard therapy that consists of Annual diethylcarbamazine (300 mg) and albendazole (400mg)
- High Dose Annual DEC/ALB: Group randomized to yearly high dose albendazole that consists of Annual diethylcarbamazine (300 mg) and albendazole (800mg)
- High Dose Semiannual DEC/ALB: Group randomized to twice-yearly high dose albendazole that consists of Annual diethylcarbamazine (300 mg) and albendazole (800mg)
Period: Overall Study
Arm/Group | Standard Therapy Annual DEC/ALB | High Dose Annual DEC/ALB | High Dose Semiannual DEC/ALB
Started | 13 | 13 | 14
Completed | 13 | 13 | 10
Not Completed | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy Annual DEC/ALB | High Dose Annual DEC/ALB | High Dose Semiannual DEC/ALB | Total
Number analyzed (Participants) | 13 | 13 | 14 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 14 | 40
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Years] | 36 [18 to 50] | 39 [18 to 50] | 37 [19 to 54] | 37 [18 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 10 | 29
  Male | 4 | 3 | 4 | 11
Region of Enrollment [Number; unit: participants]
  India | 13 | 13 | 14 | 40
Blood microfilaremia (mf/ml) [Median (Full Range); unit: MF/ML] | 412 [64 to 912] | 264 [112 to 1244] | 384 [108 to 748] | 384 [64 to 1244]

OUTCOME MEASURES:

1. Primary Outcome: Microfilarial Counts at 1 Year
Description: Night time microfilarial counts at 1 year
Time Frame: 1 year from time enrolled
Measure: Median (Full Range); unit: MF/ML
Arm/Group | Standard Therapy Annual DEC/ALB | High Dose Annual DEC/ALB | High Dose Semiannual DEC/ALB
Number analyzed (Participants) | 13 | 13 | 13
MF/ML | 0 [0 to 20] | 0 [0 to 12] | 0 [0 to 9]
Statistical Analysis 1: Comparison: Standard Therapy Annual DEC/ALB vs High Dose Annual DEC/ALB vs High Dose Semiannual DEC/ALB; Test type: Superiority or Other; p < 0.2, Fisher Exact — Adjusted for multiple comparisons

2. Secondary Outcome: Adult Worm Burdens at 2 Years
Description: Doppler detected worm nests at 2 years
Time Frame: 2 years from the time enrolled.
Population: By 2 years, 4 subjects in High Dose Group lost to followup
Measure: Median (Full Range); unit: Number of nests
Arm/Group | Standard Therapy Annual DEC/ALB | High Dose Annual DEC/ALB | High Dose Semiannual DEC/ALB
Number analyzed (Participants) | 13 | 13 | 10
Number of nests | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Standard Therapy Annual DEC/ALB vs High Dose Annual DEC/ALB vs High Dose Semiannual DEC/ALB; Test type: Superiority or Other; p = 0.9, Fisher Exact

3. Secondary Outcome: Microfilarial Levels at 2 Years
Description: Night time microfilarial levels at 2 years
Time Frame: 2 years from time enrolled
Population: By 2 years, 4 subjects in High Dose Group lost to followup
Measure: Median (Full Range); unit: MF/ML
Groups:
- Diethylcarbamazine/Albendazole -STD: Standard therapy of diethylcarbamazine (DEC) (300mg) and albendazole (400mg) yearly
  Albendazole: Comparing 400 mg to 800 mg dose
  Diethylcarbamazine: Providing diethylcarbamazine more frequently in combination with albendazole
Arm/Group | Diethylcarbamazine/Albendazole -STD | Diethylcarbamazine/Albendazole- HD1 | Diethylcarbamazine/Albendazole-HD2
Number analyzed (Participants) | 13 | 13 | 10
MF/ML | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Brugia Specific Immunoglobulin G4 (IgG4) Antibodies
Description: IgG4 antibodies directed against Brugia malayi antigen
Time Frame: 2 years
Population: By 2 years, 4 subjects in High Dose Group lost to followup
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Standard Therapy Annual DEC/ALB | High Dose Annual DEC/ALB | High Dose Semiannual DEC/ALB
Number analyzed (Participants) | 13 | 13 | 10
ng/ml | 150 [0 to 1000] | 224 [0 to 2100] | 128 [0 to 650]

ADVERSE EVENTS:
Time Frame: Every 6 months
Groups:
- High Dose Semiannual DEC/AC=LB: Group randomized to twice-yearly high dose albendazole that consists of Annual diethylcarbamazine (300 mg) and albendazole (800mg)
Arm/Group | Standard Therapy Annual DEC/ALB | High Dose Annual DEC/ALB | High Dose Semiannual DEC/AC=LB
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 9/13 | 8/13 | 11/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy Annual DEC/ALB (N=13) | High Dose Annual DEC/ALB (N=13) | High Dose Semiannual DEC/AC=LB (N=14)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 8 (8) | 11 (11)
Fever (Investigations) | 5 (5) | 4 (4) | 4 (4)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study never fully enrolled so sample size was smaller than hoped for.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No